CLINICAL TRIAL: NCT03150420
Title: A Phase 3, Intravenous Sodium Thiosulfate for Acute Calciphylaxis Treatment: A Multicenter, Randomized, Double-blind, Placebo-controlled, Clinical Trial
Brief Title: A Phase 3 Clinical Trial of Intravenous Sodium Thiosulfate in Acute Calciphylaxis Patients
Acronym: CALISTA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inability to accrue subjects that met the exclusion criterion "Any prior (within the past 30 days) or current Sodium Thiosulfate treatment".
Sponsor: Hope Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST-001
Record Dates: First submitted 2017-03-29; First posted 2017-05-12 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Calciphylaxis
Keywords: calciphylaxis; calcific uremic arteriolopathy, calcinosis; calcium metabolism disorders; metabolic diseases; sodium thiosulfate
MeSH Terms: conditions — Calciphylaxis; Calcinosis; Calcium Metabolism Disorders; Metabolic Diseases | interventions — sodium thiosulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sodium Thiosulfate (Experimental): Sodium Thiosulfate Injection (25 grams sodium thiosulfate)
  Interventions: Drug: Sodium Thiosulfate
- Placebo-Normal Saline (Placebo Comparator): 0.9% sodium chloride injection, USP (normal saline)
  Interventions: Drug: Placebo-Normal Saline

INTERVENTIONS:
Drug: Sodium Thiosulfate — Intravenous Sodium Thiosulfate Injection (25 grams sodium thiosulfate) to be administered each hemodialysis session (3 times weekly) for 3 weeks
  Other Names: Intravenous Sodium Thiosulfate Injection
  Arms: Sodium Thiosulfate
Drug: Placebo-Normal Saline — Placebo: to be administered each hemodialysis session (3 times weekly) for 3 weeks
  Other Names: 0.9% sodium chloride solution
  Arms: Placebo-Normal Saline

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled clinical trial will evaluate the efficacy and safety of intravenous Sodium Thiosulfate Injection for treatment of acute calciphylaxis-associated pain in chronic hemodialysis patients.

DETAILED DESCRIPTION:
This Phase 3, multicenter, randomized, double-blind, placebo-controlled clinical trial will evaluate the efficacy and safety of intravenous Sodium Thiosulfate Injection for treatment of acute calciphylaxis-associated pain in chronic hemodialysis patients. Acute calciphylaxis- associated pain intensity will be the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Informed of the investigational nature of the study and sign written informed consent
* Willing and able to adhere to all study-related procedures, including adherence to study medication regimen
* Male or female ≥18 years old
* End-stage renal disease on chronic hemodialysis
* Calciphylaxis with active skin lesion(s) of any morphological appearance (including but not limited to livedo, induration, ulceration, etc.) and tissue histology review consistent with calciphylaxis diagnosis. Histological features consistent with calciphylaxis will include soft tissue calcification, microthrombosis, and/or fibrointimal hyperplasia of dermal arterioles
* Acute pain associated with calciphylaxis lesions pain intensity score of ≥ 5 at initial screening on the modified BPI/SF scale
* Women of childbearing potential must have a pregnancy test (urine or serum [if anuric]) at screening and not be pregnant and willing to use an acceptable method of contraception for the entire duration of the study (3 weeks)

Exclusion Criteria:

* Peritoneal dialysis patients
* Current congestive heart failure exacerbation
* Baseline abnormalities related to QT prolongation (corrected QT interval > 470 ms), hypocalcemia (serum albumin-corrected calcium < 8 mg/dL ), metabolic acidosis (serum bicarbonate < 18 mmol/L, hypotension (resting systolic blood pressure while seated < 80), or interdialytic weight gain ≥ 4.0 kg
* History of ventricular arrhythmias including ventricular fibrillation or ventricular tachycardia associated with shortness of breath, dizziness, hypotension, or syncope
* Any prior (within the past 30 days) or current intravenous Sodium Thiosulfate Injection treatment
* Other investigational agent (drug, biologic, or device) study within the past 30 days and/or for the duration of the trial
* Pregnant or lactating women
* History of allergy to sulfites, thiosulfate, or any component in Sodium Thiosulfate Injection (sulfa allergy is not an exclusion criterion)
* Significant other acute or chronic concomitant diseases (including but not limited to hepatic, cardiovascular, pulmonary, or oncologic disease, sepsis, pulmonary edema, pulmonary embolism) that would be inconsistent with survival for at least 3 months
* Other serious concurrent or recent medical or psychiatric condition which, in the opinion of the Investigator, makes the patient unsuitable for participation in this study
* Ongoing application of dialysate admixed with iron salt e.g. ferric pyrophosphate during the entire trial period (patients who are on dialysate admixed with iron salt at screening are eligible if dialysate admixed with iron salt can be substituted with non-iron based dialysate and patients can be maintained on non-iron based dialysate therapy for the entire duration of trial period)
* Recent (within 1 week) history of surgical parathyroidectomy or scheduled for surgical parathyroidectomy during the course of the study
* History of opioid addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with 30% improvement in pain severity | randomization to 3 weeks
  To compare the effects of treatment with intravenous Sodium Thiosulfate Injection vs. placebo for the proportion of patients (responders) who achieve a ≥ 30% reduction based upon pain intensity score (modified BPI/SF).

SECONDARY OUTCOMES:
Secondary Endpoint-a: Number of patients with stabilization or improvement in calciphylaxis skin lesions. | randomization to 3 weeks
  Proportion of patients who achieve improvement or stabilization (i.e., not worsening) of skin lesions.
Secondary Endpoint-b: Occurence of surgical debridement of skin lesions and/or amputation. | during week 3
  Occurence of surgical debridement of skin lesions and/or amputation.
Secondary Endpoint-c: Occurrence of surgical debridement of skin lesions and/or amputation. | randomization to 3 weeks
  Occurrence of surgical debridement of skin lesions and/or amputation.
Secondary Endpoint-d: Time to achieve ≥ 30% improvement in pain severity | randomization to 3 weeks
  Time in days when a patient achieves a ≥ 30% improvement based upon pain intensity score (modified BPI/SF).

CONTACTS AND LOCATIONS:
Overall Officials: Craig Sherman, MD, Study Director — Hope Pharmaceuticals
Locations (21):
- United States (12):
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern University Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Veterans Administration Medical Center, Albany, New York
  - The Icahn School of Medicine at Mount Sinai Hospital, New York, New York
  - Sanford Health, Fargo, North Dakota
  - Cleveland Clinic, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Virginia Health System, Charlottesville, Virginia
  - Veterans Administration Medical Center, Salem, Virginia
- Canada (5):
  - University of Calgary Foothills Medical Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
- United Kingdom (4):
  - Salford Royal Hospital NHS Foundation Trust, Salford, Manchester
  - Hammersmith Hospital, London
  - Churchill Hospital, Oxford
  - Lister Hospital, Stevenage

IPD SHARING:
Plan to Share IPD: Undecided